CLINICAL TRIAL: NCT03646513
Title: A Safety Follow Up Study in Australian Subjects Implanted With the SMF Short Modular Femoral Stem Hip System
Status: Terminated | Type: Observational
Why Stopped: Product recalled. Sponsor decision to discontinue study.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18- 4550- 01
Record Dates: First submitted 2018-07-16; First posted 2018-08-24 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-01

CONDITIONS: Total Hip Arthroplasty (THA)
Keywords: THA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SMF Short Modular Femoral Stem Implanted Subjects: Subjects who have been implanted with the SMF Short Modular Femoral Stem for primary total hip arthroplasty.
  Interventions: Device: SMF Short Modular Femoral Hip System

INTERVENTIONS:
Device: SMF Short Modular Femoral Hip System — Primary Total Hip Arthroplasty with SMF Short Modular Femoral Stem Hip System.

SUMMARY:
This is a prospective, single arm, sequential enrolment study to collect relevant clinical and radiological data in approximately 26 subjects, at one site in Australia, who have been implanted with the SMF Short Modular Femoral Stem Hip System in a primary THA procedure to assess its safety and efficacy up to 20 years post-surgery.

DETAILED DESCRIPTION:
This is a single arm, consecutive series study to collect relevant clinical, laboratory and radiological data in up to 26 subjects, who have been implanted with the SMF Short Modular Femoral Stem THA system at 1 site in Australia.

The Baseline visit will be determined as the first visit to site after Ethics approval. This will be approximately 8-9 years post implant. Enrolled subjects will be followed up to 20 years post SMF implant.

Eligible patients will be contacted and patient status and implant revision status will be assessed at this initial contact. The subject will be given the option to participate in a prospective 12 year on-site follow-up visits for which they will provide written informed consent. Subjects who are lost to follow-up, deceased or are unwilling/unable to participate in the prospective study will be noted in the subject files and this data will be captured for analysis of study results. Data will be collected on the operative date, and implant status.

Post Baseline, the study will allow for metal ion assessments every 3 years for asymptomatic subjects and annual assessments for subjects with pain, swelling, and/or functional limitations if assessed by the Principal Investigator to be related to the SMF implant, having ruled out all other probable causes for the subject. If the subject has elevated whole blood cobalt or chromium (defined as >7ppb) a MARS MRI or CT will be obtained. These types of imaging techniques are aimed at detecting inflammatory degenerative evolution of peri articular soft tissues including pseudo-tumours. A functional Questionnaire, HOOS JR Questionnaire will be completed at all patient site visits.

Safety will be evaluated by assessing the frequency and nature of adverse events, serious adverse events and revisions.

ELIGIBILITY:
Inclusion Criteria:

* The participant has undergone primary total hip arthroplasty with the SMF short modular femoral stem at the study site and still has the original implant at the time of Ethics Committee approval of the study.
* The participant is willing and able to participate in follow-up visits at the study site.

Exclusion Criteria:

* The Subject, in the opinion of the PI, has an emotional or neurological condition that would affect their ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse.
* Subject is known to be at risk for lost to follow-up or failure to return for scheduled visits.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that have been implanted with the SMF Short Modular Femoral Stem primary stem for primary total hip arthroplasty.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen McMahon, Principal Investigator — Malabar Orthopaedic Institute, Melbourne, Australia.
Locations (1):
- Malabar Orthopaedic Clinic, Windsor, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single study site according to the study inclusion and exclusion criteria from 14 February 2019 until early termination of the study on 12 March 2020.
Pre-assignment Details: Study was prematurely terminated prior to any participants completing follow-up visits.
Period: Overall Study
Arm/Group | SMF Short Modular Femoral Stem Implanted Subjects
Started | 4
Completed | 0
Not Completed | 4
Not completed — Premature study termination | 4

BASELINE CHARACTERISTICS:
Arm/Group | SMF Short Modular Femoral Stem Implanted Subjects
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (59.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3
  Race: Asian | 1
Region of Enrollment [Number; unit: participants]
  Australia | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (28.0)

OUTCOME MEASURES:

1. Primary Outcome: Metal Ion Level
Description: All participants at Baseline and every three years afterwards up to 20 years will have whole blood collected for metal ion testing of whole blood cobalt (Co) and chromium (Cr). Symptomatic participants with pain, swelling, and/or functional limitations if assessed by the Principal Investigator to be related to the implant will have whole blood collected for metal ion testing of cobalt and chromium annually.
Time Frame: Baseline to Study Completion, up to 20 years
Population: Participants enrolled in the study with available data at the given time point for the outcome specified. Study prematurely terminated prior to any follow-up visits. Therefore, only baseline information was available.
Measure: Mean (Standard Deviation); unit: Nanomoles per litre (nmol/L)
Arm/Group | SMF Short Modular Femoral Stem Implanted Subjects
Number analyzed (Participants) | 4
Nanomoles per litre (nmol/L)
  Baseline: Cobalt (Co) | 115.0 (118.0)
  Baseline: Chromium (Cr) | 55.8 (55.5)
  20 years: Cobalt (Co): number analyzed (Participants) | 0
  20 Years: Chromium (Cr): number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Cobalt (Co) and Chromium (Cr) Metal Ions > 7 Parts-Per-Billion (Ppb)
Description: Number of participants with whole blood cobalt (Co) and/or chromium (Cr) > 7 ppb (Yes/No). Participants as 'Yes' to Co and/or Cr will have Metal Artifact Reduction Sequence (MARS) Magnetic Resonance Imaging (MRI) performed (or Computerized tomography (CT) if MRI is contraindicated). This is used to detect pseudotumors, abductor muscle atrophy, and tendinous pathology in patients with painful metal-on-metal (MOM) hip arthroplasty.
Time Frame: Baseline to study completion, up to 20 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SMF Short Modular Femoral Stem Implanted Subjects
Number analyzed (Participants) | 4
Participants
  Baseline: Cobalt (Co): Yes | 2
  Baseline: Cobalt (Co): No | 2
  Baseline: Chromium (Cr): Yes | 0
  Baseline: Chromium (Cr): No | 4
  20 Years: Cobalt (Co): number analyzed (Participants) | 0
  20 Years: Chromium (Cr): number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Short Modular Femoral (SMF) Stem Revision
Description: Number of participants with a revision of any component of the SMF Short Modular Femoral Stem for any reason as a result of an adverse event. Revisions captured at any time during the study duration (up to 20 years) from the point of informed consent signing.
Time Frame: Study Completion, up to 20 years
Population: Study prematurely terminated prior to any follow-up visits.
Arm/Group | SMF Short Modular Femoral Stem Implanted Subjects
Number analyzed (Participants) | 0

4. Secondary Outcome: Radiographic Assessment: Loosening
Description: Standard of Care Radiographic Assessment for loosening indicated by radiolucencies > 2 millimeters (mm). In a cemented arthroplasty, this lucency at the bone-cement interface indicates the formation of a fibrous membrane (representing the lucency). Periprosthetic lucencies wider than 2 mm and/or progressive lucencies are signs of abnormality.
Time Frame: Baseline to study completion, up to 20 years
Population: Study prematurely terminated prior to any follow-up visits.
Arm/Group | SMF Short Modular Femoral Stem Implanted Subjects
Number analyzed (Participants) | 0

5. Secondary Outcome: Radiographic Assessments: Surface Wear
Description: Number of participants with evidence of surface wear (Yes/No) as indicated by early osteolysis, implant migration, or other clinical or radiographic abnormalities such as pseudo tumors or corrosion.
Time Frame: Baseline to study completion, up to 20 years
Population: Study prematurely terminated prior to any follow-up visits.
Arm/Group | SMF Short Modular Femoral Stem Implanted Subjects
Number analyzed (Participants) | 0

6. Secondary Outcome: The Hip Osteoarthritis Outcomes Score Junior (HOOS JR) Questionnaire
Description: The HOOS JR. questionnaire consists of 6 questions. These focus on 3 categories: joint pain, stiffness and function in daily living. The HOOS JR. questionnaire, allows patients to rate each activity by indicating the amount of pain or disability they experience while carrying them out. Raw scores are added up and then converted to an interval score (0-100) using an interval table. The final interval score represents a patients total joint disability where 0 corresponds to total joint disability (i.e., worse outcome) and 100 is perfect joint health (i.e., best outcome).
Time Frame: Baseline to study completion, up to 20 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMF Short Modular Femoral Stem Implanted Subjects
Number analyzed (Participants) | 4
score on a scale
  Baseline | 100 (0)
  20 Years: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected for all participants enrolled in the study to early termination of the study, approximately 1 year.
Description: All participants enrolled in the study were evaluated for adverse events (AEs) from 14 February 2019 to premature termination of the study on 12 March 2020. At each contact with the participant, the Investigator sought information on AEs by specific questioning and, as appropriate, by assessment of the participant.
Arm/Group | SMF Short Modular Femoral Stem Implanted Subjects
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
The study was prematurely termination by the Sponsor with a limited number of enrolled participants. Only preoperative (baseline) participant data was available because no participant completed any follow-up visits due to early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03646513/Prot_SAP_000.pdf